CLINICAL TRIAL: NCT01946620
Title: A Randomised, Double-blind, Double Dummy, Parallel Group Study Comparing Fluticasone Propionate / Formoterol Fumarate (Flutiform®) 250/10 µg (2 Puffs BID) and Flutiform® 125/5 µg (2 Puffs BID) Versus Formoterol Fumarate Dihydrate (Atimos®) 12 µg (1 Puff BID) in Subjects With Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: A Study to Show That Flutiform is Well Tolerated and Effective in the Treatment of COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FLT3509; 2012-004162-17 (EudraCT Number)
Record Dates: First submitted 2013-09-10; First posted 2013-09-19 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Exacerbations; FEV1 ≤ 50%
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — fluticasone-formoterol; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Flutiform 250/10 micrograms (Experimental): Flutiform 250/10 µg (2 puffs twice daily)
  Interventions: Drug: Flutiform
- Flutiform 125/5 micrograms (Experimental): Flutiform 125/5 µg (2 puffs twice daily)
  Interventions: Drug: Flutiform
- Formoterol 12 micrograms (Active Comparator): Formoterol 12 µg 1 puff twice daily
  Interventions: Drug: Formoterol

INTERVENTIONS:
Drug: Flutiform
  Arms: Flutiform 125/5 micrograms; Flutiform 250/10 micrograms
Drug: Formoterol
  Arms: Formoterol 12 micrograms

SUMMARY:
Efficacy of Fluticasone/Formoterol in COPD Treatment. The Effect study.

DETAILED DESCRIPTION:
This study is a multi-centre, randomised, double-blind, active-controlled, parallel-group study, in male and female subjects who will be assigned into 1 of 3 treatment groups based on 1:1:1 ratio. Following a 2 week run-in phase all subjects will receive treatment for 1 year (52 weeks) followed by a final follow up 2 weeks after their last visit, during this time subjects will be required to attend 10 clinic visits while the final follow up can be completed by telephone. Throughout the study subjects will be assessed on a mixture of symptom based measurements as well as lung function tests to monitor their progress in the study.

ELIGIBILITY:
Inclusion:

1. Male or Female subjects aged ≥ 40 years at screening visit:

   1. Female subjects of child bearing potential (less than 1 year post-menopausal) must have a negative urine pregnancy test prior to first dose of study medication, be non-lactating, and willing to use adequate and highly effective methods of birth control throughout the study such as sterilisation, implants, injectables, combined oral contraceptives, some intra-uterine devices, sexual abstinence or vasectomised partner.
   2. Male subjects with a partner of child bearing potential must be willing to use adequate and highly effective methods of birth control throughout the study
2. Smoking history of ≥10 packs per year.
3. Diagnosis of COPD
4. History of ≥ moderate or severe COPD exacerbations in previous year.
5. Willing and able to replace current COPD therapy with study medication.
6. Able to demonstrate correct use of a pMDI without a spacer.
7. Willing and able to attend all study visits and complete study assessments.
8. Able to provide signed informed consent.

Exclusion:

1. Ongoing moderate or severe exacerbation of COPD (see section 10)
2. Current diagnosis of asthma
3. Documented evidence of α1-antitrypsin deficiency as the underlying cause of COPD
4. Other active respiratory disease such as active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung disease, cystic fibrosis, bronchiolitis obliterans
5. Previous lung resection
6. Use of long-term oxygen therapy (LTOT) at least 12 hours daily or mechanical ventilation
7. Chest X-ray or CT scan that reveals evidence of clinically significant abnormalities reflective of active disease not believed to be due to COPD
8. Evidence of uncontrolled cardiovascular disease
9. Evidence of clinically significant renal, hepatic, gastrointestinal, or psychiatric disease
10. Current malignancy or a previous history of cancer which has been in remission for < 5 years (basal cell or squamous cell carcinoma of the skin which has been resected is not excluded)
11. Clinically significant sleep apnoea requiring use of continuous positive airway pressure (CPAP) device or non-invasive positive pressure ventilation (NIPPV) device
12. Participation in the acute phase of a pulmonary rehabilitation programme within 4 weeks prior to screening or during the study
13. Known or suspected history of drug or alcohol abuse in the last 2 years
14. Requiring treatment with any of the prohibited concomitant medications
15. Known or suspected hypersensitivity or contraindication to any of the study drugs or excipients
16. Received an investigational drug within 30 days of the screening visit (12 weeks if an oral or injectable steroid).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1767 (Actual)
Dates: Start 2013-10; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Annual rate of moderate and severe COPD exacerbations | 52 weeks
  To show superiority in the efficacy of flutiform 250/10 µg (2 puffs BID) compared with formoterol 12 µg (1 puff BID) based on the annual rate of moderate and severe COPD exacerbations

SECONDARY OUTCOMES:
Annual rate of moderate and severe COPD exacerbations | 52 Weeks
  To show superiority in the efficacy of flutiform 125/5 µg (2 puffs BID) compared with formoterol 12 µg (1 puff BID) based on the annual rate of moderate and severe COPD exacerbations. (Different dose to Primary Outcome)
Efficacy confirmed by lack of exacerbations, lung function and safety by collection of adverse events in all patients throughout the study. | 52 Weeks
  To compare flutiform (at each dose) with formoterol 12 µg (1 puff BID) for the secondary efficacy, and safety endpoints.

CONTACTS AND LOCATIONS:
Locations (15):
- Sofia, Bulgaria
- Hamburg, Germany
- Budapest, Hungary
- Riga, Latvia
- Vilnius, Lithuania
- Skopje, North Macedonia
- Trzemeszno Lubuskie, Poland
- Bacau, Romania
- Moscow, Russia
- Prešov, Slovakia
- Cape Town, South Africa
- Gyeonggido, South Korea
- Barcelona, Spain
- Kyiv, Ukraine
- London, United Kingdom

REFERENCES:
- See also: Link to Results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=FLT3509